CLINICAL TRIAL: NCT04074850
Title: The Long-term Consequences After Traumatic Brain Injury in the Elderly: a Prospective Study
Brief Title: The Long-term Consequences After Traumatic Brain Injury in the Elderly
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62848
Record Dates: First submitted 2019-07-25; First posted 2019-08-30 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-11

CONDITIONS: Traumatic Brain Injury; Aging; Cognitive Impairment; Quality of Life
Keywords: Traumatic Brain Injury; Elderly; Cognitive Impairment; Quality of life; Impact; Health care economic costs
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TBI group: A cohort of patients admitted to UZ Leuven from 1999 to 2019 due to Traumatic Brain Injury and fulfilling our inclusion and exclusion criteria will be recruited.
  Inclusion criteria will be: ≥ 65 years old at the time of the accident, admitted to UZ Leuven from 1999 and 2019, all injury severities, classified by the Glasgow Coma Scale (GCS) (mild (GCS 13-15), moderate (GCS 9-12) or severe (GCS ≤8)), and having signed the informed consent to participate in the study.
  Exclusion criteria will be: < 65 years old, admitted to UZ Leuven in a different period from 1999-2019, diagnosis of other neurodegenerative diseases before the TBI, cognitive and motor disturbances caused by any other pathology before the TBI, previous alcohol/drugs abuse, and not having signed the informed consent to participate in the study.

SUMMARY:
A better understanding of the injury patterns, injury severity, risk profiles, consequences and impact of Traumatic Brain Injury (TBI) in the elderly population is necessary due to the increasing incidence and prevalence of TBI in this population and its high economic impact on society. Therefore, this study aims at describing the long-term consequences of TBI. In order to achieve that goal, injury patterns, injury severity and risk profiles for TBI in the elderly will be mapped. Moreover, a retrospective assessment of brain damage, co-morbidities and post-traumatic history, and a prospective assessment of cognitive functions and quality of life in a 20 years range after TBI will be performed. Finally, a statistical correlation of TBI and different types of neurodegenerative diseases, and an economic costs analysis will be done. All the obtained results will be used to develop a new prognostic tool for the course of the outcomes of TBI in the elderly population.

DETAILED DESCRIPTION:
A database of over 1200 patients will be created by the retrospective capture of the following data in UZ Leuven database:

Injury mechanisms data:

In order to create a map of injury patterns, severity and criteria that allow for identifying which accident circumstances ageing adults should reasonably be protected against, including a kinematics tolerance curve for the elderly brain that can be used for protection purposes, a retrospective analysis of data related to injury mechanisms, registered in the patient's clinical records, will be performed for the cohort of patients.

Clinical data:

Data regarding the following parameters will be retrospectively collected in UZ Leuven database for the studty cohort: age, sex, cause of injury, GCS, pupillary reactivity, hypoxia, hypotension, hypothermia and Marshall CT classification at the time of admission. Moreover, Glasgow Outcome Scale (GOSE) at 6 months after the accident, obtained in the context of routine clinical practice, will also be considered.

These data will be correlated with the results obtained during the injury patterns, injury severity and risk profiles mapping, in order to better understand what accident types are most risky to eventually result in poor outcome.

Economic data:

In order to know what is the economic impact that TBI in the elderly has on society, hospital costs for the clinical management in the study cohort will be retrospectively extracted from the financial database of UZ Leuven.

All these data will be anonymized and no informed consent will be used in this part of the study.

Current status assessment:

In this part of the project, all the patients ≥65 years old admitted to UZ Leuven due to TBI between 1999 and 2019, and fulfilling previously explained inclusion and exclusion criteria, will be contacted through a phone call by an investigator of this project, and offered to participate in the study.

UZ Leuven administration (MIR) has access to a central national database, so the list of patients will be screened prior to the start of the phone calls in order to exclude the patients that are deceased and avoid calling them.

The informed consent form will be distributed among the patients via post or e-mail, depending on their preferences. Patients will have to send the signed informed consent form back to the researchers via post or e-mail in order to be assessed.

Once the researchers receive the signed informed consent form, patients will be called again and they will have the cognitive and quality of life evaluation, which consists of:

-Cognitive evaluation: the Telephone Interview for Cognitive Status (TICS) tool will be used to study cognitive functions in the cohort. It is a 11-items screening test for cognitive functions, including word list memory, orientation, attention, repetition, conceptual knowledge and nonverbal praxis. The necessary time to perform it is 10 min or less.

Moreover, the patients' level of education will be asked, registered and correlated with clinical data, cognitive functions and quality of life outcomes.

* Sleep quality assessment: the sleep quality in our cohort will be assessed using the Pittsburgh Sleep Quality Index.
* Quality of life evaluation: the Quality of Life after Brain Injury (QOLIBRI) tool will be used to assess the quality of life in the cohort. It is a 37-item questionnaire with six subscales that measure quality of life in the domains of cognition, self, daily life and autonomy, social relationships, emotions, and physical problems. The approximate time necessary to fill this questionnaire in is 10 min.

Once the investigators get the signed informed consent, injury mechanisms data, clinical data and clinical-care related economic data will be collected from UZ Leuven database and correlated to the cognitive, sleep quality and quality of life outcomes. Also, for all the patients in the study cohort that live in the surrounding areas of Leuven and have UZ Leuven as a reference hospital after TBI, a retrospective revision of the clinical records will be performed for the identification of diagnosis for neurodegenerative diseases that developed after TBI.

Based on previous statistical figures, the investigators expect to have a cohort of over 500 patients for this current status assessment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old at the time of the accident
* admitted to UZ Leuven from 1999 and 2019
* all injury severities
* classified by the Glasgow Coma Scale (GCS) (mild (GCS 13-15), moderate (GCS 9-12) or severe (GCS ≤8))
* having signed the informed consent to participate in the study.

Exclusion Criteria:

* < 65 years old
* admitted to UZ Leuven in a different period from 1999-2019
* diagnosis of other neurodegenerative diseases before the TBI
* cognitive and motor disturbances caused by any other pathology before the TBI
* previous alcohol/drugs abuse
* not having signed the informed consent to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 65 years old with a Traumatic Brain Injury diagnose that were admitted in UZ Leuven after the accident between 1999 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Injury mechanisms evaluation | August 2019-June 2021
  Injury mechanisms will be studied in order to better understand which accident circumstances ageing adults should reasonably be protected against. Results will be included in a descriptive report.
Economic cost evaluation | August 2019-June 2021
  In order to know what is the economic impact that TBI in the elderly has on society, hospital costs for the clinical management in our cohort will be retrospectively extracted from the financial database of UZ Leuven.
Cognitive functions assessment | August 2019-November 2022
  A telephonic cognitive evaluation will be performed using the Telephone Interview for Cognitive Status (TICS) tool, which is a 11-items screening test for cognitive functions, including word list memory, orientation, attention, repetition, conceptual knowledge and nonverbal praxis. The TICS total score has a maximum of 41 points and higher scores mean better cognitive outcomes. The necessary time to perform it is 10 min or less.
  Moreover, the patients' level of education will be asked, registered and correlated with clinical data, cognitive functions and quality of life outcomes.
Quality of life assessment | August 2019-November 2022
  A telephonic quality of life evaluation will be performed using the Quality of Life after Brain Injury (QOLIBRI) tool, which is a 37-item questionnaire with six subscales that measure quality of life in the domains of cognition, self, daily life and autonomy, social relationships, emotions, and physical problems.The QOLIBRI scores are reported on a 0-100 scale, where 0=worst possible quality of life and 100=best possible quality of life. The approximate time necessary to fill this questionnaire in is 10 min.
Sleep quality assessment | August 2020-November 2022
  A telephonic sleep quality assessment will be performed using the Pittsburgh Sleep Quality Index. In this scale, seven component scores are derived, each scored from 0 (which means no difficulty) to 3 (severe difficulty). The global score ranges between 0 and 21 points. Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium